CLINICAL TRIAL: NCT07007429
Title: Effects of Stimulated Occlusal Imbalance and Jaw Clenching on Balance and Fall Risk in Stroke Patients
Brief Title: Effects of Occlusal Imbalance and Clenching on Balance in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEUFTR-9
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator and the researcher administering intervention will be different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ipsilesional Side Stimulated Occlusal Imbalance Group (Experimental): In this group, occlusal imbalance will be induced by placing a cotton roll on the ipsilesional occlusal surfaces of the patients.
  Interventions: Other: Ipsilesional Side Stimulated Occlusal Imbalance
- Contralesional Side Stimulated Occlusal Imbalance Group (Experimental): In this group, occlusal imbalance will be induced by placing a cotton roll on the contralesional occlusal surfaces of the patients.
  Interventions: Other: Contralesional Side Stimulated Occlusal Imbalance
- Bilateral Cotton Roll with Jaw Clenching Group (Experimental): Patients in the bilateral cotton roll with jaw clenching group will clench their teeth while cotton rolls are placed on both sides of the occlusal surfaces.
  Interventions: Other: Bilateral Cotton Roll with Jaw Clenching

INTERVENTIONS:
Other: Ipsilesional Side Stimulated Occlusal Imbalance — In this group, a 1 cm thick cotton roll will be placed on the ipsilesional occlusal surfaces of the patients, and they will be instructed to hold it in place without clenching.
  Arms: Ipsilesional Side Stimulated Occlusal Imbalance Group
Other: Contralesional Side Stimulated Occlusal Imbalance — In this group, a 1 cm thick cotton roll will be placed on the contralesional occlusal surfaces of the patients, and they will be instructed to hold it in place without clenching.
  Arms: Contralesional Side Stimulated Occlusal Imbalance Group
Other: Bilateral Cotton Roll with Jaw Clenching — In this group, a 1 cm thick cotton roll will be placed on both occlusal surfaces, and the patients will then be instructed to clench their teeth.
  Arms: Bilateral Cotton Roll with Jaw Clenching Group

SUMMARY:
The aim of the study is to investigate the effects of stimulated occlusal imbalance and jaw clenching on balance and fall risk in patients with stroke.

DETAILED DESCRIPTION:
This randomized controlled study will be conducted on a minimum of 42 stroke patients who meet the inclusion and exclusion criteria. Patients included in the study will be randomly assigned to one of three groups: the ipsilateral side stimulated occlusal imbalance group, the contralateral side stimulated occlusal imbalance group, or the bilateral jaw clenching group.

ELIGIBILITY:
Inclusion Criteria:

* Having chronic stroke,
* A Mini-Mental State Examination score of 24 or higher,
* Being between 18 and 75 years of age,
* Having a Brunnstrom stage of 4 or above,
* Ability to stand independently for 20 seconds or more,
* Ability to walk independently for 10 meters, using assistive devices or orthoses if necessary,
* Having opposing mandibular and maxillary second premolars or first molars

Exclusion Criteria:

* The presence of severe osteoarthritis in the lower extremity,
* The presence of cancer or diabetic neuropathy,
* The presence of vestibular disorder,
* The presence of lower extremity ulceration or amputation,
* Hemodynamic instability,
* The presence of other neurological disorders (such as multiple sclerosis, Parkinson's disease),
* Having experienced an acute lower extremity injury in the last six weeks,
* History of lower extremity surgery,
* Alcohol consumption in the last 24 hours
* Posterior circulation stroke involving the basilar artery or cerebellum

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Overall Postural Stability Index Measurement | Change from baseline overall postural stability index immediately after the intervention
  This index will be assessed by measuring deviations of the center of gravity in the anteroposterior and mediolateral directions. Lower scores indicate smaller deviations and better postural stability. The test will be performed on a stable platform with two trials of 30 seconds each. The average of the two trials will be automatically calculated by the TechnoBody balance system.
Fall Risk Assessment | Change from baseline fall risk immediately after the intervention
  Fall risk will be assessed by measuring the patient's ability to maintain balance on an unstable platform. Based on their ability to maintain balance, a fall risk score will be generated, with higher scores indicating a greater risk of falling. The test will be performed with two 30-second trials. The average of the two trials will be calculated automatically by the TechnoBody balance system.

SECONDARY OUTCOMES:
Anteroposterior Stability Index Measurement | Change from baseline anteroposterior stability index immediately after the intervention
  The anteroposterior stability index will be assessed by measuring deviations of the center of gravity in the anteroposterior direction. Lower scores indicate smaller deviations and better anteroposterior postural stability. The test will be performed on a stable platform with two trials of 30 seconds each. The average of the two trials will be automatically calculated by the TechnoBody balance system.
Mediolateral Stability Index Measurement | Change from baseline mediolateral stability index immediately after the intervention
  The mediolateral stability index will be assessed by measuring deviations of the center of gravity in the mediolateral direction. Lower scores indicate smaller deviations and better mediolateral postural stability. The test will be performed on a stable platform with two trials of 30 seconds each. The average of the two trials will be automatically calculated by the TechnoBody balance system.
Weight Bearing Distribution Assessment | Change from baseline weight bearing distribution immediately after the intervention
  Weight-bearing distribution will be assessed by measuring the percentage of body weight borne by each limb during quiet standing. Lower asymmetry values indicate more balanced weight distribution and better postural stability. The test will be performed on a stable platform with two trials of 30 seconds each. The average of the two trials will be automatically calculated by the TechnoBody balance system.

CONTACTS AND LOCATIONS:
Overall Officials: ömer dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; burak mavuş, M.Sc., Principal Investigator — Bolu Abant İzzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital
Locations (1):
- Bolu İzzet Baysal Fizik Tedavi ve Rehabilitasyon Eğitim ve Araştırma Hastanesi, Bolu, Merkez, Turkey (Türkiye)

REFERENCES:
- [Background] Arene N, Hidler J. Understanding motor impairment in the paretic lower limb after a stroke: a review of the literature. Top Stroke Rehabil. 2009 Sep-Oct;16(5):346-56. doi: 10.1310/tsr1605-346. PMID 19903653
- [Background] Lamb SE, Ferrucci L, Volapto S, Fried LP, Guralnik JM; Women's Health and Aging Study. Risk factors for falling in home-dwelling older women with stroke: the Women's Health and Aging Study. Stroke. 2003 Feb;34(2):494-501. PMID 12574566
- [Background] Tyson SF, Hanley M, Chillala J, Selley A, Tallis RC. Balance disability after stroke. Phys Ther. 2006 Jan;86(1):30-8. doi: 10.1093/ptj/86.1.30. PMID 16386060
- [Background] Yates JS, Lai SM, Duncan PW, Studenski S. Falls in community-dwelling stroke survivors: an accumulated impairments model. J Rehabil Res Dev. 2002 May-Jun;39(3):385-94. PMID 12173758
- [Background] Divani AA, Vazquez G, Barrett AM, Asadollahi M, Luft AR. Risk factors associated with injury attributable to falling among elderly population with history of stroke. Stroke. 2009 Oct;40(10):3286-92. doi: 10.1161/STROKEAHA.109.559195. Epub 2009 Jul 23. PMID 19628798
- [Background] Tecco S, Polimeni A, Saccucci M, Festa F. Postural loads during walking after an imbalance of occlusion created with unilateral cotton rolls. BMC Res Notes. 2010 May 25;3:141. doi: 10.1186/1756-0500-3-141. PMID 20500818
- [Background] Tecco S, Salini V, Calvisi V, Colucci C, Orso CA, Festa F, D'Attilio M. Effects of anterior cruciate ligament (ACL) injury on postural control and muscle activity of head, neck and trunk muscles. J Oral Rehabil. 2006 Aug;33(8):576-87. doi: 10.1111/j.1365-2842.2005.01592.x. PMID 16856955
- [Background] Fujimoto M, Hayakawa L, Hirano S, Watanabe I. Changes in gait stability induced by alteration of mandibular position. J Med Dent Sci. 2001 Dec;48(4):131-6. PMID 12160250
- [Background] Asseman F, Gahery Y. Effect of head position and visual condition on balance control in inverted stance. Neurosci Lett. 2005 Feb 28;375(2):134-7. doi: 10.1016/j.neulet.2004.10.085. Epub 2004 Nov 24. PMID 15670656
- [Background] Giannakopoulos NN, Schindler HJ, Hellmann D. Co-contraction behaviour of masticatory and neck muscles during tooth grinding. J Oral Rehabil. 2018 Jul;45(7):504-511. doi: 10.1111/joor.12646. Epub 2018 May 30. PMID 29761534
- [Background] Giannakopoulos NN, Schindler HJ, Rammelsberg P, Eberhard L, Schmitter M, Hellmann D. Co-activation of jaw and neck muscles during submaximum clenching in the supine position. Arch Oral Biol. 2013 Dec;58(12):1751-60. doi: 10.1016/j.archoralbio.2013.09.002. Epub 2013 Sep 20. PMID 24200301
- [Background] Giannakopoulos NN, Hellmann D, Schmitter M, Kruger B, Hauser T, Schindler HJ. Neuromuscular interaction of jaw and neck muscles during jaw clenching. J Orofac Pain. 2013 Winter;27(1):61-71. doi: 10.11607/jop.915. PMID 23424721